CLINICAL TRIAL: NCT03354364
Title: Efficacy of Pea Hull Fiber Supplementation on Gastrointestinal Transit Time-induced Reduction in Proteolytic Fermentation and Enhancement of Wellness in Individuals With Lifestyle-related Chronic Disease and Overweight. (Phase 3)
Brief Title: Efficacy of Pea Hull Fiber in Chronic Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Saskatchewan Pulse Growers (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: IRB201701457
Record Dates: First submitted 2017-11-21; First posted 2017-11-27 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Kidney Disease, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Receives pea hull fiber snack for the first 4 weeks and then control snack for the last 4 weeks of the study with 4-week washout between them.
  Interventions: Dietary Supplement: Pea hull fiber; Dietary Supplement: Control
- Group 2 (Active Comparator): Receives control snack for the first 4 weeks and then pea hull fiber snack for the last 4 weeks of the study with 4-week washout between them
  Interventions: Dietary Supplement: Pea hull fiber; Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Pea hull fiber — Snacks containing 15 g/day of ground pea hulls.
Dietary Supplement: Control — Snacks without added fiber.

SUMMARY:
The purpose of this study is to determine the effects of daily consumption of snacks with and without pea hull fiber on gastrointestinal function, gastrointestinal symptoms, food intake, appetite, changes in fecal and microbial composition and activity. Fifty maintenance hemodialysis hemodialysis and CKD patients in stage 4 or 5 will be recruited to participate in a randomized, blinded, 13-week cross-over study evaluating snack foods containing 15 g/d of pea hull fiber.

DETAILED DESCRIPTION:
Maintenance hemodialysis hemodialysis and CKD patients in stage 4 or 5 (n=50) will be recruited for the study. A randomized, controlled, double-blind, cross-over study will be carried out. Following a 1-week baseline, participants will be assigned to receive snacks with pea hull fiber or control followed by a 4-week wash-out period, and then crossed over to the second intervention. Snacks with added pea hull fiber (15 g/d) and control will be provided to participants in identical packaging. Participants will collect 4 days of stools during the baseline week, week 5, 9, and 13 and analyzed for mineral content. Microbiota composition will be analyzed including microbial diversity, qPCR to quantify changes and 16S rRNA sequencing to identify pea hull fiber effects on specific bacteria. Following baseline, participants will attend a second visit and anthropometric and demographic information will be collected and we will measure blood pressure, the body composition by bioelectrical impedance analysis (BIA), and handgrip strength using a dynamometer.

Throughout the study, participants must complete a daily questionnaire to evaluate the transit time (eg. Bristol Stool Scale), stool frequency, and compliance. Every week, questionnaires to evaluate appetite (eg. SNAQ) and GI wellness (eg. GSRS - Gastrointestinal Symptom Response Scale) will be administered. During each study visit, participants will complete a questionnaire to evaluate the quality of life. In addition, the dietary data (24-hour diet recalls) will be collected by phone during the baseline week and during the last week of each period. During baseline, treatment and each washout, fasting blood will be collected and analyzed for a comprehensive metabolic panel with eGFR, in addition to microbial metabolites (e.g., indoxyl sulfate and p-cresyl sulfate), and inflammatory markers (e.g. CRP, TNFα, IL-6).

ELIGIBILITY:
Inclusion Criteria:

* 18-85 years of age.
* Kidney disease stage 4 or 5 (including dialysis).
* Willing and able to complete the Consent Form in English.
* Willing to have height, weight, blood pressure, handgrip strength, and body composition measured and provide demographic information (e.g. age, race, sex).
* Willing to consume pea hull fiber snack or control snack for a 56-day period, 28 day for each type of snack.
* Willing to complete a daily, and weekly, and monthly questionnaires regarding appetite, wellness, and transit time, and quality of life throughout the entire 13-week study.
* Willing to provide three 24-hr diet recalls by phone during baseline and last week of each period.
* Willing to provide 16 days of stools and 4 blood samples throughout the study.

Exclusion Criteria:

* Do not meet the above criteria.
* Have known gastrointestinal disease (i.e., inflammatory bowel disease, malignancy, celiac disease), previous colorectal surgery.
* Allergies to ingredients in study foods provided.
* Are pregnant or lactating

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-08-19 (Actual)

PRIMARY OUTCOMES:
Uremic molecule - p-cresyl sulfate | baseline, 5 weeks, 9 weeks, 13 weeks
  Change in serum levels of microbial metabolic product, p-cresyl sulfate

SECONDARY OUTCOMES:
Uremic molecules (various) | baseline, 5 weeks, 9 weeks, 13 weeks
  Change in serum levels microbial metabolic products (e.g. indoxyl sulfate, TMAO, phenylacetyl glutamine etc.)
Fecal content of metabolites and minerals | at baseline, week 5, week 9 and week 12.
  Change in fecal concentration of microbial metabolites and minerals
Number of stools per week | 13 weeks
  Change in number of stools per week and mean number of stools per week per period
Stool form rating | 13 weeks
  Change in stool form determined using Bristol Stool Form Scale
Gastrointestinal symptom score | at weeks 1 through 13
  Change in gastrointestinal symptom score determined by GSRS (Gastrointestinal Symptom Response Scale)
Fecal microbiota profile changes | baseline, weeks 5, 9 and 13
  change at phylum and genus levels; changes in operational taxonomic units (OTUs)
Dietary intake | baseline, weeks 5, 9 and 13
  Change in dietary energy, macronutrient and fiber intake
Appetite | at weeks 1 through 13
  Change in appetite determined by SNAQ questionnaire
Quality of Life | baseline, weeks 5, 9 and 13
  Change in Kidney Disease Quality of Life questionnaire (KDQOL®-36)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy J Dahl, PhD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - Village of Gainesville, Gainesville, Florida
  - Food Science and Human Department, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: Undecided